CLINICAL TRIAL: NCT03368352
Title: Effects of Melatonin on Sleep, Ventilatory Control and Cognition at Altitude.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Naomi Deacon, Research Scholar, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 170200
Record Dates: First submitted 2017-11-20; First posted 2017-12-11 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Altitude Hypoxia; Ventilation; Sleep; Oxidative Stress; Neurocognitive Dysfunction
Keywords: Melatonin; Altitude; Sleep; Ventilation; Cognition
MeSH Terms: conditions — Altitude Sickness; Respiratory Aspiration; Cognition Disorders | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Normoxia (No Intervention): Sleep in normal room air with no drug
- Hypoxia with Placebo (Placebo Comparator): Sleep in hypoxic tent after taking Placebo 1 hour before bed.
  Interventions: Other: Hypoxia
- Hypoxia with Melatonin (Experimental): Sleep in hypoxic tent after taking 5 mg Melatonin before bed.
  Interventions: Dietary Supplement: Melatonin

INTERVENTIONS:
Dietary Supplement: Melatonin — Dietary supplement melatonin
  Arms: Hypoxia with Melatonin
Other: Hypoxia — Sleep in a hypoxic tent simulating high altitude
  Arms: Hypoxia with Placebo

SUMMARY:
Low oxygen at altitude causes pauses in breathing during sleep, called central sleep apnea. Central sleep apnea causes repeated awakenings and poor sleep. Low oxygen itself and the induced oxidative stress can damage mental function which is likely worsened by poor sleep. Reduced mental function due to low oxygen can pose a serious danger to mountain climbers. However there is also mounting evidence that even in populations of people that live at high altitudes and are considered adapted, low oxygen contributes to reductions in learning and memory. Therefore there is a serious need for treatments which may improve sleep, control of breathing and mental function during low oxygen. Melatonin is a hormone produced in the brain during the night which regulates sleep patterns with strong antioxidant and anti-inflammatory properties. A study previously reported that melatonin taken 90 mins before bed at 4,300 m (14,200 ft) induced sleep earlier, reduced awakenings and improved mental performance the following day. However how melatonin caused these effects was not determined. Therefore this study aims to determine how melatonin effects control of breathing, sleep and mental performance during exposure to low oxygen.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Sleep disorders
* Pregnant females
* Smokers (quit ≥ 1 year ago acceptable)
* Any known cardiac (apart from treated hypertension with acceptable drugs, see below), pulmonary (including asthma), renal, neurologic (including epilepsy), neuromuscular, hepatic disease, or patients with diabetes.
* Prior or current use of melatonin.
* Use of any medications that may affect sleep or breathing, blood-thinning medications (anticoagulants), antioxidants, anti-inflammatories, medications that suppress the immune system (immunosuppressants), diabetes medications and birth control pills.
* A psychiatric disorder, other than mild depression; e.g. schizophrenia, bipolar disorder, major depression, panic or anxiety disorders.
* Substantial alcohol (>3oz/day) or use of illicit drugs.
* Previous occurrence of high altitude pulmonary or cerebral edema.
* Recent exposure to altitude (>8000ft) in the last month or having slept at an altitude >6000ft in the last month.
* Inability to provide written informed consent or able to complete the experiment.
* Non-English speakers (necessary to complete neurocognitive testing).
* More than 10 cups of beverages with caffeine (coffee, tea, soda/pop) per day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Neurocognitive function | 30 minutes after arousal from sleep
  Stroop-color word test median number of errors. Higher numbers indicate worse performance.
Endothelial function | 5 minutes after arousal from sleep
  Reactive hypermedia index via EndoPat
Lipid peroxidation in serum | immediately after arousal from sleep
  Concentration of Malondialdehyde in serum samples
Hypercapnic hypoxic ventilatory sensitivity | 1 hour after arousal from sleep
  This is the one outcome. It is the gain of the ventilatory response to changes in CO2, during sustained hypoxia. Delta minute ventilation / delta mmHg CO2 during sustained hypoxia

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Sleep Lab, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No